CLINICAL TRIAL: NCT04206007
Title: The Safety and Feasibility of UMC119-06 Cell Therapy in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Mesenchymal Stem Cells for The Treatment of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meridigen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMC119-06-COPD-01
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-12

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UMC119-06 (Experimental): Human Umbilical Cord Derived-Mesenchymal Stem Cells, Single treatment by intravenous infusion.
  Interventions: Biological: UMC119-06

INTERVENTIONS:
Biological: UMC119-06 — Cohort 1: Low does of UMC119-06 Cohort 2: Medium does of UMC119- 06 Cohort 3: High does of UMC119-06

SUMMARY:
The clinical study with UMC119-06 is designed to investigate the safety in patients with Chronic Obstructive Pulmonary Disease. This will be a dose escalation, open label, single-center study in adult with chronic obstructive pulmonary disease. UMC119-06 is ex vivo cultured human umbilical cord tissue-derived mesenchymal stem cells product which is intended for treatment of chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a leading cause of morbidity and mortality worldwide, predicted to be the third leading cause of death in adults by 2020. Patients with COPD are characterized with airflow limitation and chronic inflammation, which is caused by cigarette smoking, noxious particles or gases. These inhaled irritants will induce inflammation, emphysema and fibrosis though chronic exposure. The current pharmacological treatment of COPD is symptomatic and is mainly based on bronchodilators, such as selective β2-adrenergic agonists (short-and long-acting), anticholinergics, theophylline, or a combination of these drugs. In patients with continuing exacerbations, inhaled corticosteroids (ICSs) may be added in the form of a triple fixed dose combination inhaler that includes ICSs, long-acting β2-agonists (LABA) and inhaled long-acting muscarinic antagonists (LAMA). Although current clinical treatment strategies can improve and stabilize COPD states and quality of life, none of them are able to modify the progressive decline in lung function which is the hallmark of this disease. Therefore, development of new therapeutic modalities to improve the clinical outcomes and prognosis of COPD in adult patients is of urgent need. Among the more innovative, experimental therapies, mesenchymal stromal cells (MSCs) are proposed as a novel therapy with potential in treatment of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of age between ≥ 40 through ≤ 75 years.
* Subjects with diagnosis of COPD based on the Global Initiative for Chronic Obstructive Lung Diseases (GOLD) standard.
* Subjects with a post-bronchodilator FEV1/FVC ratio <0.7.
* Subjects with a post-bronchodilator FEV1 % predicted value ≥ 50% and < 80%.
* Subjects with score ≥ 2 in the modified Medical Research Council Dyspnea Scale (mMRC).
* Subjects with in COPD Assessment Test (CAT) score ≥ 10.
* Subjects with body weight between 40 to 90 kg.
* Subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided.
* Women of child-bearing potential should have a negative urine pregnancy test prior to administration of investigational product, UNLESS they meet the following criteria:

  1. Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40 mIU/m, OR;
  2. 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy
* If a male and heterosexually active with a female of childbearing potential, the subject must agree to use a double barrier method of birth control (or must have been surgically sterilized) and to not donate sperm during the study.

Exclusion Criteria:

* Subjects with history of any type of malignancy.
* Subjects with major surgery (body organs that require anesthesia, such as tumor removal, open chest, heart surgery, abdominal surgery, intracranial surgery, or normal surgery for more than 3 hours, etc.) within previous 30 days.
* Subjects who are pregnant (or plan to become pregnant within 3 months of investigational product treatment) or lactating.
* Subjects who have a significant concomitant illness as judged by principal investigator (PI).
* Subjects with known human immunodeficiency virus infection or who are immune compromised.
* Subjects with a known history of alcohol abuse or drug abuse within the 5 years before study treatment administration.
* Subjects who are current smokers.
* Subjects unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation.
* Subjects with a history of severe allergic or anaphylactic reactions.
* Subjects with known allergy or hypersensitivity to any component of the formulation or hypersensitivity to any component of the formulation (normal saline and human serum albumin).
* Subjects who have participated in another clinical study of new investigational therapies or have received an investigational therapy within the 12 weeks before study drug administration.
* Subjects with known Alpha-1 antitrypsin deficiency.
* Subjects with current active infection including pulmonary infection, systemic infection or severe local infections.
* Subjects with exacerbation of COPD within the 12 weeks before study treatment administration.
* Subjects who have the following conditions in laboratory tests at screening;

  1. >2 × upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST); or
  2. >2 × ULN for serum creatinine.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of adverse events related to administration of UMC119-06. | 3 months from the day of administration
  * Incidence of Treatment-Emergent Adverse Events (TEAEs).
  * Incidence of withdrawals due to Adverse Events(AEs).

SECONDARY OUTCOMES:
Changes in Forced Vital Capacity (FVC). | 15 months from the day of administration.
  Improvement in clinical function as assessed by mean change in Forced Vital Capacity (FVC).
Changes in Forced Expiratory Volume in One Second (FEV1). | 15 months from the day of administration.
  Improvement in clinical function as assessed by mean change in Forced Expiratory Volume in One Second (FEV1).
Changes in the ratio of Forced Expiratory Volume in One Second to the Forced Vital Capacity (FEV1/FVC). | 15 months from the day of administration
  Improvement in clinical function as assessed by mean change in the ratio of Forced Expiratory Volume in One Second to the Forced Vital Capacity (FEV1/FVC).
Changes in exercise performance using 6-min walk test (6MWT). | 15 months from the day of administration.
  Improvement in clinical function as assessed by mean change in exercise performance using 6-min walk test (6MWT).
Changes in Quality Of Life using St. George's Respiratory Questionnaire Safety (SGRQ). | 15 months from the day of administration.
  Scores range from 0 (no impairment) to 100 (maximum impairment), with higher scores indicating more limitation. A decrease in score represents a decrease in disease related symptoms. Improvement in clinical function as assessed by mean change in Quality Of Life using St. George's Respiratory Questionnaire Safety (SGRQ).
Changes in modified medical research council (mMRC) -dyspnea scale. | 15 months from the day of administration.
  Scores range from 0 (no dyspnea) to 4 (severe dyspnea), with higher scores indicate worse COPD control. Improvement in clinical function as assessed by mean change in modified medical research council (mMRC) -dyspnea scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare., New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No